CLINICAL TRIAL: NCT01296022
Title: Randomized Trial to Study the Efficacy and Adverse Effects of the Subcutaneous and Transvenous Implantable Cardioverter Defibrillator (ICD) in Patients With a Class I or IIa Indication for ICD Without an Indication for Pacing
Brief Title: A PRospective, rAndomizEd Comparison of subcuTaneOous and tRansvenous ImplANtable Cardioverter Defibrillator Therapy
Acronym: PRAETORIAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, R.E. Knops, Drs. R.E. Knops, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL34725.018.10; NL34725.018.10 (Other: Centrale Commissie Mensgebonden Onderzoek)
Record Dates: First submitted 2011-01-12; First posted 2011-02-15 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Ventricular Arrhythmias
Keywords: Heart rhythm disturbances; Implantable cardiac defibrillator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subcutaneous ICD (Active Comparator): Subcutaneous Implantable Cardioverter Defibrillator
  Interventions: Device: Implantation of subcutaneous ICD
- Transvenous ICD (Active Comparator): Transvenous Implantable Cardioverter Defibrillator
  Interventions: Device: Implantation of transvenous ICD

INTERVENTIONS:
Device: Implantation of subcutaneous ICD — Implantation of subcutaneous ICD
  Arms: Subcutaneous ICD
Device: Implantation of transvenous ICD — Implantation of transvenous ICD
  Arms: Transvenous ICD

SUMMARY:
This randomized controlled trial will outline the advantages and disadvantages of the subcutaneous implantable cardioverter defibrillator (ICD) compared to the transvenous ICD.

DETAILED DESCRIPTION:
Background of the study: The use of implantable cardioverter defibrillators (ICDs) is an established therapy for the prevention of death from ventricular arrhythmia. Recently a new subcutaneous ICD has been introduced, eliminating the need for transvenous lead placement in or on the heart which is mandatory in the transvenous ICD. The new subcutaneous ICD therapy already proved to be feasible and safe and is an approved therapy in Europe. It is likely that the eliminated need for transvenous lead placement substantially reduces the implantation related complications and elongates lead longevity and thus reduces inappropriate shocks associated with lead fractures. On the other hand it is unclear whether the lack of capability to provide antitachy-pacing (ATP) in the subcutaneous ICD may be a limitation for patients with frequent recurrent ventricular tachycardia. This randomized controlled trial will outline the advantages and disadvantages of the subcutaneous ICD.

Objectives of the study: (1) To compare the subcutaneous ICD to the transvenous ICD for major adverse events (i.e. inappropriate shocks, acute and chronic implant related complications and lead- or device related complications). (2) To determine to which degree the lack of ATP function leads to more appropriate shocks in patients with a subcutaneous ICD.

Study design: Multicenter, prospective, randomized controlled trial with either treatment with the transvenous ICD or subcutaneous ICD (1:1).

Study population: 2x425 patients with class I or IIa indication for ICD therapy without an indication for pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Patients with class I or IIa indication for ICD therapy according to the ACC/AHA/ESC 2006 Guidelines for Management of Patients With Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death

Exclusion Criteria:

* Patients with documented therapy refractory monomorphic ventricular tachycardia
* Patients having an indication for pacing therapy
* Patients with ventricular tachycardia less than 170 bpm
* Patients failing appropriate QRS/T-wave sensing with the S-ICD ECG patient screening tool provided by Cameron Health/Boston Scientific
* Patients with incessant ventricular tachycardia
* Patients with a serious known concomitant disease with a life expectancy of less than one year
* Patients with circumstances that prevent follow-up (no permanent home or address, transient, etc.)
* Patients who have had a previous ICD implant
* Patient who receive cardiac contractility modulation therapy or are likely to receive cardiac contractility modulation therapy.
* Patients who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with implantable cardioverter defibrillator (ICD) related adverse events | 48 months
  ICD related adverse events are defined as inappropriate shocks and/or implant-, lead- and device related complications. An inappropriate shock is shock therapy for anything else but ventricular fibrillation or ventricular tachycardia. Implant related complications are defined as ICD related infections, ICD related bleedings, thrombotic events, need for lead reposition, post-implant pneumothorax, post-implant hematothorax, or post-implant perforation/tamponade. Lead- or device related complications are all complications related to the lead or device.

SECONDARY OUTCOMES:
Number of Major Adverse Cardiac Event (MACE) | 48 months
  MACE is defined as cardiac death, myocardial infarction, percutaneous coronary intervention, coronary artery bypass grafting and/or any valve surgery
Number of appropriate shocks | 48 months
  An appropriate shock is shock therapy for ventricular fibrillation or ventricular tachycardia.
Number of inappropriate shocks | 48 months
  Inappropriate shocks are defined as above.
Number of complications individually | 48 months
  Complications are defined as above.
Quality of life | 30 months
  The quality of life is measured by the SF-36 and Duke Activity Status Index questionnaires.
Time to successful therapy | 48 months
  Time to successful therapy is the time between the start of VT or VF until the first successful shock or first successful ATP episode. This includes the time of sensing and charging.
First shock conversion efficacy | 48 months
  First shock conversion efficacy is the amount of patients with VT or VF who are successfully converted with the first shock given by the transvenous ICD or subcutaneous ICD.
Implant procedure time | 48 months
  Implant procedure time is the time between the first incision and placement of the last suture (skin-to-skin time).
Hospitalization rate | 48 months
  The hospitalization rate is the number of days a patient is admitted to the hospital associated with ICD implantation.
Fluoroscopy time | 48 months
  Fluoroscopy time is the total time that fluoroscopy is used during the implantation of either the transvenous ICD or subcutaneous ICD.
Cardiac (pre-)syncope events | 48 months
  Cardiac syncope is a loss of consciousness due to cerebral hypoperfusion caused by cardiac arrhythmias or presumed cardiac arrhythmias
Cross-overs to the other arm | 48 months
  A crossover to the other arm is defined as a patient who for any reason after randomization is switched to the other ICD arm
Cardiac decompensation | 48 months
  Cardiac decompensation refers to acute failure of the heart to maintain adequate blood circulation for which hospitalization and medical treatment is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Reinoud E Knops, MD, PhD, Principal Investigator — Academic Medical Center - University of Amsterdam (AMC-UvA); Arthur A.M. Wilde, MD, PhD, Study Chair — Academic Medical Center - University of Amsterdam (AMC-UvA)
Locations (39):
- United States (10):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Mount SinaÏ Hospital, New York, New York
  - Columbia University, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
- Na Homolce Hospital, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- Germany (7):
  - Herzzentrum Dresden, Dresden
  - Universitätsklinikum Jena, Jena
  - Universtätsklinikum Kiel, Kiel
  - Herzzentrum Leipzig, Leipzig
  - Universitätsklinikum Mannheim, Mannheim
  - University Hospital Grosshadern, Munich
  - Universitätsklinikum Wurzburg, Würzburg
- Netherlands (14):
  - Noordwest Hospital, Alkmaar
  - Flevoziekenhuis, Almere Stad
  - Academic Medical Center - University of Amsterdam (AMC-UvA), Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - VU Medical Center, Amsterdam
  - Amphia Hospital, Breda
  - Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Maastricht University Medical Center, Maastricht
  - St. Antonius Hospital, Nieuwegein
  - Radboudumc, Nijmegen
  - ErasmusMC, Rotterdam
  - Isala Klinikum Zwolle, Zwolle
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Heart & Chest Hospital, Liverpool
  - Hammersmith Hospital, London
  - Saint Bartholomew's Hospital, London
  - St. Georges Hospital of London, London
  - Oxford University Hospitals NHS Trust, Oxford

REFERENCES:
- [Background] Olde Nordkamp LR, Knops RE, Bardy GH, Blaauw Y, Boersma LV, Bos JS, Delnoy PP, van Dessel PF, Driessen AH, de Groot JR, Herrman JP, Jordaens LJ, Kooiman KM, Maass AH, Meine M, Mizusawa Y, Molhoek SG, van Opstal J, Tijssen JG, Wilde AA. Rationale and design of the PRAETORIAN trial: a Prospective, RAndomizEd comparison of subcuTaneOus and tRansvenous ImplANtable cardioverter-defibrillator therapy. Am Heart J. 2012 May;163(5):753-760.e2. doi: 10.1016/j.ahj.2012.02.012. PMID 22607851
- [Result] Knops RE, Olde Nordkamp LRA, Delnoy PHM, Boersma LVA, Kuschyk J, El-Chami MF, Bonnemeier H, Behr ER, Brouwer TF, Kaab S, Mittal S, Quast ABE, Smeding L, van der Stuijt W, de Weger A, de Wilde KC, Bijsterveld NR, Richter S, Brouwer MA, de Groot JR, Kooiman KM, Lambiase PD, Neuzil P, Vernooy K, Alings M, Betts TR, Bracke FALE, Burke MC, de Jong JSSG, Wright DJ, Tijssen JGP, Wilde AAM; PRAETORIAN Investigators. Subcutaneous or Transvenous Defibrillator Therapy. N Engl J Med. 2020 Aug 6;383(6):526-536. doi: 10.1056/NEJMoa1915932. PMID 32757521
- [Result] Knops RE, van der Stuijt W, Delnoy PPHM, Boersma LVA, Kuschyk J, El-Chami MF, Bonnemeier H, Behr ER, Brouwer TF, Kaab S, Mittal S, Quast ABE, Smeding L, Tijssen JGP, Bijsterveld NR, Richter S, Brouwer MA, de Groot JR, Kooiman KM, Lambiase PD, Neuzil P, Vernooy K, Alings M, Betts TR, Bracke FALE, Burke MC, de Jong JSSG, Wright DJ, Jansen WPJ, Whinnet ZI, Nordbeck P, Knaut M, Philbert BT, van Opstal JM, Chicos AB, Allaart CP, Borger van der Burg AE, Clancy JF, Dizon JM, Miller MA, Nemirovsky D, Surber R, Upadhyay GA, Weiss R, de Weger A, Wilde AAM, Olde Nordkamp LRA; PRAETORIAN Investigatorsdouble dagger. Efficacy and Safety of Appropriate Shocks and Antitachycardia Pacing in Transvenous and Subcutaneous Implantable Defibrillators: Analysis of All Appropriate Therapy in the PRAETORIAN Trial. Circulation. 2022 Feb;145(5):321-329. doi: 10.1161/CIRCULATIONAHA.121.057816. Epub 2021 Nov 14. PMID 34779221
- [Result] Knops RE, Pepplinkhuizen S, Delnoy PPHM, Boersma LVA, Kuschyk J, El-Chami MF, Bonnemeier H, Behr ER, Brouwer TF, Kaab S, Mittal S, Quast ABE, van der Stuijt W, Smeding L, de Veld JA, Tijssen JGP, Bijsterveld NR, Richter S, Brouwer MA, de Groot JR, Kooiman KM, Lambiase PD, Neuzil P, Vernooy K, Alings M, Betts TR, Bracke FALE, Burke MC, de Jong JSSG, Wright DJ, Jansen WPJ, Whinnett ZI, Nordbeck P, Knaut M, Philbert BT, van Opstal JM, Chicos AB, Allaart CP, Borger van der Burg AE, Dizon JM, Miller MA, Nemirovsky D, Surber R, Upadhyay GA, Weiss R, de Weger A, Wilde AAM, Olde Nordkamp LRA. Device-related complications in subcutaneous versus transvenous ICD: a secondary analysis of the PRAETORIAN trial. Eur Heart J. 2022 Dec 14;43(47):4872-4883. doi: 10.1093/eurheartj/ehac496. PMID 36030464
- [Derived] Olde Nordkamp LRA, de Veld JA, Ghani A, Kuschyk J, Bonnemeier H, Bode K, Boersma LVA, de Weger A, de Jong JSSG, Jansen WPJ, Alings M, Bijsterveld N, El-Chami MF, Beukema RJ, Vernooy K, Philbert BT, Neuzil P, Nordbeck P, van Opstal JM, Allaart CP, Wright DJ, Knaut M, Betts TR, Whinnett ZI, Lambiase PD, de Groot JR, Chicos AB, Nemirovksy D, Kaab S, Mittal S, Borger van der Burg AE, Dijkshoorn LA, Pepplinkhuizen S, van der Stuijt W, Dizon JM, Miller MA, Behr ER, Burke MC, Kooiman KM, Quast ABE, Brouwer TF, Wilde AAM, Smeding L, Knops RE; PRAETORIAN-XL Investigators. Device-Related Complications in Transvenous Versus Subcutaneous Defibrillator Therapy During Long-Term Follow-Up: The PRAETORIAN-XL Trial. Circulation. 2025 Jul 22;152(3):172-182. doi: 10.1161/CIRCULATIONAHA.125.074576. Epub 2025 Apr 25. PMID 40279654
- [Derived] Olde Nordkamp LRA, Pepplinkhuizen S, Ghani A, Boersma LVA, Kuschyk J, El-Chami MF, Behr ER, Brouwer TF, Kaab S, Mittal S, Quast ABE, van der Stuijt W, Smeding L, de Veld JA, Tijssen JGP, Bijsterveld NR, Richter S, Brouwer MA, de Groot JR, Kooiman KM, Lambiase PD, Neuzil P, Vernooy K, Alings M, Betts TR, Bracke FALE, Burke MC, de Jong JSSG, Wright DJ, Jansen WPJ, Whinnett ZI, Nordbeck P, Knaut M, Philbert BT, van Opstal JM, Chicos AB, Allaart CP, Borger van der Burg AE, Dizon JM, Miller MA, Nemirovsky D, Surber R, Upadhyay GA, Weiss R, de Weger A, Wilde AAM, Knops RE; PRAETORIAN Investigators. Inappropriate Therapy and Shock Rates Between the Subcutaneous and Transvenous Implantable Cardiac Defibrillator: A Secondary Analysis of the PRAETORIAN Trial. Circ Arrhythm Electrophysiol. 2024 Dec;17(12):e012836. doi: 10.1161/CIRCEP.124.012836. Epub 2024 Dec 3. PMID 39624908
- [Derived] Knops RE, de Veld JA, Ghani A, Boersma LVA, Kuschyk J, El Chami MF, Bonnemeier H, Behr ER, Brouwer TF, Kaab S, Mittal S, Pepplinkhuizen S, Quast ABE, Smeding L, van der Stuijt W, de Weger A, Bijsterveld NR, Richter S, Brouwer MA, de Groot JR, Kooiman KM, Lambiase PD, Neuzil P, Vernooy K, Alings M, Betts TR, Bracke FALE, Burke MC, de Jong JSSG, Wright DJ, Jansen WPJ, Whinnett ZI, Nordbeck P, Knaut M, Philbert BT, van Opstal JM, Chicos AB, Allaart CP, Borger van der Burg AE, Dizon JM, Miller MA, Nemirovksy D, Surber R, Upadhyay GA, Tijssen JGP, Wilde AAM, Olde Nordkamp LRA; PRAETORIAN Investigators. Quality of Life in Subcutaneous or Transvenous Implantable Cardioverter-Defibrillator Patients: A Secondary Analysis of the PRAETORIAN Trial. Circ Cardiovasc Qual Outcomes. 2024 Nov;17(11):e010822. doi: 10.1161/CIRCOUTCOMES.124.010822. Epub 2024 Nov 19. PMID 39561235